CLINICAL TRIAL: NCT03181295
Title: Screening While You Wait: A Technology-based Intervention to Facilitate Actionable Exercise Prescriptions in Primary Care
Brief Title: Screening While You Wait: An Intervention to Facilitate Exercise in Primary Care
Acronym: SWYW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2016-0126-B
Record Dates: First submitted 2017-05-16; First posted 2017-06-08 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Physical Activity
Keywords: Family Medicine; Primary Care; Exercise prescriptions; Technology
MeSH Terms: conditions — Motor Activity | interventions — Health Resources

STUDY DESIGN:
Intervention Model Description: Single-centre, pilot step wedge trial, with graduated, random intervention roll-out across the clinical setting in four steps
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Standard periodic health review (PHR) appointment. [As patients will get a survey about PA levels prior to their PHR, this may affect their likelihood of addressing PA during their PHR.]
- Usual care plus intervention (Experimental): Standard PHR appointment plus personalized exercise Rx and resources
  Interventions: Behavioral: Personalized exercise Rx and resources

INTERVENTIONS:
Behavioral: Personalized exercise Rx and resources — Patients will receive the IPAQ to collect baseline PA levels as well as questions evaluating precursors to behaviour change and identifying medical conditions that may affect PA capability. In the Electronic Medical Record chart, a 'stamp' will be automatically created, accompanied by a link which will open a printable 'toolkit' with individualized PA recommendations, a personalized exercise Rx, as well as educational and community resources, all based on the patient's survey responses. The exercise Rx and resources can be edited by the PCP based on the resulting discussion between patient and PCP, and printed during the PHR for the patient to take home. The exercise Rx and resources will also be emailed to the patient following their appointment.
  Arms: Usual care plus intervention

SUMMARY:
Despite knowing that exercise improves health, primary care providers (PCPs) do not regularly assess physical activity (PA) levels or use proven techniques to help patients to increase their PA levels. Studies have shown that PCPs don't talk to patients about their PA levels because they don't feel they have adequate knowledge or resources to help their patients. Additionally they don't feel they have time to provide personalized advice regarding PA.

This study will use tablet computers and email to engage patients in contemplating their own PA levels and starting conversations with their PCPs. Electronic surveys delivered via tablets and email prior to periodic health reviews will be used to support customized, patient-centred health care. The patient's survey responses will be used to develop a printable 'toolkit' with individualized PA recommendations, a personalized exercise prescription (Rx), as well as patient-specific educational and community resources. The exercise Rx and resources can be edited by the PCP based on the resulting discussion between patient and PCP.

The overarching aim of this study is to determine how the use of technology in family doctors' offices can help patients to engage with their PCPs regarding PA and ultimately increase their PA levels.

DETAILED DESCRIPTION:
The study will take place at the academic Women's College Hospital (WCH) Family Practice (FP) in Toronto, Canada. The clinic provides over 50,000 patient visits per year and is split into four sub-teams for operational purposes. These teams have unique members with no crossover of PCPs. Patients typically see their own PCP for planned care visit (e.g., preventative care and chronic disease management) but access any PCP available when more acute issues arise.

The PA surveys are administered via Ocean by CognisantMD. Ocean connects patients, PCPs, and researchers using secure surveys on tablets in the FP waiting room and online patient surveys that integrate with WCH FP Electronic Medical Records.

This is a pilot step wedge trial, with graduated, random intervention roll-out across the clinical setting in four steps over five time intervals. Eligible patients presenting to the clinic during the study period will be allocated to intervention or control depending on whether the PCP they have booked to see has had the intervention 'turned-on'. The order determining when each PCP and his or her team change from control to intervention is randomly assigned. This design was chosen to avoid the risk of intervention contamination and to enable logistics of implementation. The teams will receive the control and intervention according to the following schedule:

Time Interval 1: Team A-D Control Time Interval 2: Team A Intervention, Team B-D Control Time Interval 3: Team A+B Intervention, Team C+D Control Time Interval 4: Team A-C Intervention, Team D Control Time Interval 5: Team A-D Intervention

ELIGIBILITY:
Family physicians (and the patients they care for) are eligible for the study if they are active staff at WCH FP and have consented to participating.

Participating family physicians will assist in identifying potential participants and confirm that patients are appropriate participants for a study of this nature.

Patient inclusion criteria:

* Adult WCH FP patients aged 18-79
* Attending a PHR - formerly known as a 'complete physical' examination

Patient exclusion criteria:

* Non-English speaking patients (due to inability to translate the study materials at the pilot-phase)
* Patients with dementia or cognitive impairment (due to the burden of completing survey materials potentially outweighing the uncertain benefit of intervention)
* Patients who have a major ongoing illness (due to the possibility of their injury/illness interfering with their PA capabilities)
* Patients who are pregnant (due to limitations in modifying PA level between baseline and follow-up)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Metabolic Equivalent of Task-minutes per week | 4 months post-intervention
  The primary outcome will assess intervention effectiveness in terms of total PA; specifically, Metabolic Equivalent of Task (MET)-minutes per week will be calculated from the International Physical Activity Questionnaire (IPAQ).

SECONDARY OUTCOMES:
Measures of motivation (based on the Health Action Process Approach) | 4 months post-intervention
  Assessed in both intervention and control patients
Measures of self-efficacy (based on the Health Action Process Approach) | 4 months post-intervention
  Assessed in both intervention and control patients
Proportion of eligible patients providing outcome data | 4 months post-intervention
  Assessed in both intervention and control patients
Proportion of eligible patients provided the exercise Rx | 0-2 weeks post-intervention
  Intervention patients only
Estimated time spent on PA | 0-2 weeks post-intervention
  Intervention patients only
Satisfaction with PA advice | 0-2 weeks post-intervention
  Intervention patients only

CONTACTS AND LOCATIONS:
Overall Officials: Noah Ivers, Principal Investigator — Family Doctor and Research Scientist
Locations (1):
- Women's College Hospital Family Practice, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwarzer R. Modeling health behavior change: How to predict and modify the adoption and maintenance of health behaviors. Applied Psychology 2008 Jan;57(1):1-29.
- [Background] Lippke S, Ziegelmann JP, Schwarzer R. Stage-specific adoption and maintenance of physical activity: testing a three-stage model. Psychology of Sport and Exercise. 6 (5): 585-603, 2005.
- [Background] Lippke S, Ziegelmann JP, Schwarzer R. Initiation and Maintenance of Physical Exercise: Stage-Specific Effects of a Planning Intervention. Research in Sports Medicine 12: 221-240, 2004.
- [Background] Lippke S, Schwarzer R, Ziegelmann JP, Scholz U, Schuz B. Testing stage-specific effects of a stage-matched intervention: a randomized controlled trial targeting physical exercise and its predictors. Health Educ Behav. 2010 Aug;37(4):533-46. doi: 10.1177/1090198109359386. Epub 2010 Jun 14. PMID 20547760
- [Background] Schwarzer R, Lippke S, Luszczynska A. Mechanisms of health behavior change in persons with chronic illness or disability: the Health Action Process Approach (HAPA). Rehabil Psychol. 2011 Aug;56(3):161-70. doi: 10.1037/a0024509. PMID 21767036
- [Derived] Agarwal P, Kithulegoda N, Bouck Z, Bosiak B, Birnbaum I, Reddeman L, Steiner L, Altman L, Mawson R, Propp R, Thornton J, Ivers N. Feasibility of an Electronic Health Tool to Promote Physical Activity in Primary Care: Pilot Cluster Randomized Controlled Trial. J Med Internet Res. 2020 Feb 14;22(2):e15424. doi: 10.2196/15424. PMID 32130122